CLINICAL TRIAL: NCT06752967
Title: Hormonal Control of Energy and Macronutrient Intake in Obesity
Brief Title: Hormonal Control of Energy and Macronutrient Intake in Obesity (MEMORY)
Acronym: MEMORY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Novo Nordisk A/S (Industry); University of Leeds (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-24048302
Record Dates: First submitted 2024-11-05; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Normal Weight; Overweight
Keywords: ad libitum buffet; Food preferences; Macronutrient; Appetite; Appetite hormones; FGF21; Glucagon
MeSH Terms: conditions — Obesity; Overweight; Food Preferences

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protein liquid test meal (Experimental): Liquid test meal high in protein.
  Interventions: Other: High protein liquid test meal
- Carbohydrate liquid test meal (Experimental): Liquid test meal high in carbohydrates.
  Interventions: Other: High carbohydrate liquid test meal

INTERVENTIONS:
Other: High protein liquid test meal — High protein liquid test meal consisting of whey protein, water and sugar-free coadial mix for flavour.
  Arms: Protein liquid test meal
Other: High carbohydrate liquid test meal — High carbohydrate liquid test meal consisting of sucrose, water and sugar-free coadial mix for flavour.
  Arms: Carbohydrate liquid test meal

SUMMARY:
The overall aim of the MEMORY study is to examine the concept of 'food memory' - how specific macronutrient compositions influence subsequent food preference and intake, and whether this differs across the BMI range from normal weight to obesity.

DETAILED DESCRIPTION:
45 people (age 18-45 years old) with normal weight (BMI between 18.5-24.9 kg/m^2, n=15), overweight (BMI between 25-29.9 kg/m^2, n=15), and obesity (BMI above 30 kg/m^2, n=15) will participate in this randomized cross-over study. Participants will complete one screening visit and two test visits.

During their test visits participants will be served a liquid meal consisting of either carbohydrate (sucrose) or protein (whey protein) diluted in water and sugar-free cordial mix for flavor. Participants will be served either carbohydrate or protein at their first visit and the opposite at their second visit in random order. The test visits will include clinical assessment (body weight, body composition, and blood pressure); Blood samples; Visual analogue scales for assessment of subjective appetite; Ad libitum buffet for assessment of energy intake. Participants will complete the Steno Biometric Food Preference Task (SBFPT), a computerized task measuring food choice, explicit liking, and implicit and explicit wanting with concomitant biometric measurements.

Time: -60 minutes (fasting), 0 minutes (liquid test meal), 150 minutes (ad libitum test buffet).

Descriptive data will be collected at the screening visit and will include body weight (kg); BMI, kg/m^2; Fasting blood samples; Urine sample (future research); Adipose tissue biopsy (future research). Participants will also answer questionnaires regarding Socioeconomic status (SES), Control over eating (CoEQ), Health and wellbeing (SF-36), physical activity (international physical activity ((IPAQ)), and chronotype (morningsness/eveningsness ((MEQ)).

The specific research aims are:

1. To investigate whether intake of high-sucrose or high-protein affects subsequent food sensory-specific preference and different food intake from an ad libitum buffet, and whether this differs between individuals across the BMI range from normal weight to obesity.
2. To investigate whether the plasma FGF21 and glucagon responses:

   1. Differ between the above-mentioned macronutrient compositions,
   2. Are associated to subsequent food sensory-specific preference and macronutrient intake from an ad libitum buffet, and
   3. Differ between individuals across the BMI range from normal weight to obesity.
3. To investigate whether the postprandial responses of well-known appetite-related hormones, as well as unexplored metabolites and proteins:

   1. Differ between the above-mentioned macronutrient compositions,
   2. Are associated to subsequent food sensory-specific preference and macronutrient intake from an ad libitum buffet, and
   3. Differ between individuals across the BMI range from normal weight.
4. To identify new biomarkers facilitating patient stratification and optimize future treatment of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* For women: Regular menstruation
* BMI-range 18.5-39.9 kg/m^2

Exclusion Criteria:

* Not able or willing to eat or drink the test meals because of e.g., allergy or intolerance
* Daily smoking
* For women: Pregnancy / planned pregnancy (within the study period) / lactating
* Self-reported history of an eating disorder
* Self-reported weight change (kg) within two months prior to inclusion
* HbA1c ≥48 mmol/mol
* Treatment with antidepressants
* Alcohol/drug abuse or in treatment with disulfiram (antabus) at time of inclusion
* Uncontrolled medical issues including but not limited to cardiovascular pulmonary, rheumatologic, hematologic, oncologic, infectious, gastrointestinal, or psychiatric disease; diabetes or other endocrine disease; immunosuppression
* Current treatment with medication which significantly affect appetite or energy balance (e.g., GLP-1 receptor agonists)
* Bariatric surgery
* Unable to understand the informed consent and the study procedures
* Concomitant participation in intervention studies
* Participant's withdrawal of the informed consent
* Other safety concerns - judged by the investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in energy intake from sweet tasting carbohydrates. | Measured after meal consumption at t=150 min
  The difference in energy intake (E%) from sweet tasting carbohydrates during the ad libitum buffet in response to the high carbohydrate vs. high protein isocaloric liquid test meals.

SECONDARY OUTCOMES:
Difference in self-reported energy intake | Measured 24-hours after test visits
  Difference in 24-h self-reported energy intake (KJ) from carbohydrate, protein, and fat and total energy intake in response to the high carbohydrate vs. high protein isocaloric liquid meals.
Difference in energy intake from fat | Measured after meal consumption at t=150 min
  Difference in energy intake (KJ) from protein during the ad libitum buffet in response to the high carbohydrate vs. high protein isocaloric liquid meals.
Difference in energy intake from sweet tasting carbohydrates. | Measured after meal consumption at t=150 min
  The difference in energy intake (KJ) from sweet tasting carbohydrates during the ad libitum buffet in response to the high carbohydrate vs. high protein isocaloric liquid test meals.
Difference in energy intake from protein | Measured after meal consumption at t=150 min
  Difference in energy intake (KJ) from protein during the ad libitum buffet in response to the high carbohydrate vs. high protein isocaloric liquid meals.
Food choice | Measured during test visits (T=-60 min and T=120 min)
  Food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT. Food choice is determined based on frequency of selection made within each food category. The scores range from 0-48 i.e. 0 = foods within a specific food category have not been selected at all to 48 = foods within a specific food category have been selected 48 times.
Food attention | Measured during test visits (T=-60 min and T=120 min)
  Measured using eye tracking in response to looking at food pictures during SBFPT.
  Includes the following parameters: Gaze: Time spent (ms and %) andrevisits (n); and fixations: Time to first fixation (ms), time spent (ms and %), fixation count (n), first fixation duration (ms), average fixation duration (ms). Distance to screen (mm), and gaze direction bias (ratio) which is calculated as the number of trials in which the first fixation was directed to a food image as a proportion to all trials. A bias score ˃0.5 indicates attention towards one food image, a bias score equal to 0.5 indicates no bias, and a bias score <0.5 indicates attention towards the other food images.
Food reaction time | Measured during test visits (T=-60 min and T=120 min)
  Reaction time during forced food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fatsavoury and low-fat sweet foods) examined from the SBFPT.
Explicit liking | Measured during test visits (T=-60 min and T=120 min)
  Explicit liking of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT. Explicit liking is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how pleasant would it be to taste this foodright now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Implicit wanting | Measured during test visits (T=-60 min and T=120 min)
  Implicit wanting of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT. Implicit wanting is assessed based on food choice and response time for selected and non-selected food items as well as mean response time (a frequency-weighted algorithm).
  In this frequency-weighted algorithm a positive score indicates a morerapid preference for a food type over another food type and a negative score indicates the opposite. A score of zero indicates that food types are equally preferred. The frequency weighted algorithm isused so the implicit wanting score is influenced by both selection (positively contributing to the score) and non-selection (negatively contributing to the score) of food type. Scores for implicit wanting typically range from -100-100 (due to reaction time there is no fixedmin-max value)
Explicit wanting | Measured during test visits (T=-60 min and T=120 min)
  Explicit wanting of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT. Explicit wanting is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how much do you want some of this food now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Unspecified exploratory outcome | Measured during test visits (T=-60 min and T=120 min)
  Unspecified exploratory outcomes related to the 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT.
Subjective appetite sensations | Measured at specific time points during test visits (fasted, T=15 min, T=30 min, T=60 min, T= 75 min, T=90 min, T=105 min, T=120 min, T=150 min)
  Rated using visual analogue scales and includes sensations of: Hunger, fullness, satiety, prospective food consumption, wellbeing, nausea, thirst, desire to eat meat, salty, or sweet. The scale range is 0-100 mm and each end represent the extremes e.g. hunger rating: "I am not hungry at all" to "I have never been this hungry before".
Difference in plasma FGF21 | Measured during screening visit and test visit (fasted, T=15 min, T=30 min, T=60 min, T= 75 min, T=90 min, T=105 min, T=120 min, T=150 min)
  Difference in plasma FGF21 concentrations in response to the high carbohydrate vs. high protein isocaloric liquid meals.
Difference in plasma glucagon levels | Measured during screening visit and test visit (fasted, T=15 min, T=30 min, T=60 min, T= 75 min, T=90 min, T=105 min, T=120 min, T=150 min)
  Difference in plasma glucagon levels in response to the high carbohydrate vs. high protein isocaloric liquid meals.
Metabolites | Measured at fasted state (LDL/HDL, cholesterol, triglycerides, FFA) and to T=15 min, T=30 min, T=60 min, T= 75 min, T=90 min, T=105 min, T=120 min, T=150 min (glucose, FFA)
  Concentrations of metabolites including but not limited to: glucose, triglycerides, cholesterol (LDL/HDL), Free-Fatty Acids (FFA) in response to the high carbohydrate vs. high protein isocaloric liquid meals.
Hormones | Measured during screening visit and test visit (fasted, T=15 min, T=30 min, T=60 min, T= 75 min, T=90 min, T=105 min, T=120 min, T=150 min)
  Concentrations of hormones related to regulation of appetite, glucose and lipid metabolism (including but not limited to: Insulin, glucagon, ghrelin, Glucagon-Like Peptide-1 (GLP-1), Glucose-Dependent Insulinotropic polypeptide (GIP), C-peptide, Peptide YY (PYY),Fibroblast Growth Factor 21 (FGF21), Growth Differentiation Factor 15 (GDF15), Leptin, Cholecystokinin (CCK), Pancreatic Peptide (PP).
Biomarkers | Measured during screening visit and test visit (fasted, T=15 min, T=30 min, T=60 min, T= 75 min, T=90 min, T=105 min, T=120 min, T=150 min)
  Circulating biomarkers measured with metabolomics, lipidomics, proteomics
Electrolytes | Measured during test visits (fasted, T=15 min, T=30 min, T=60 min, T= 75 min, T=90 min, T=105 min, T=120 min, T=150 min)
  Concentrations of electrolytes including but not limited to: Natrium and Kalium
Inflammatory markers | Measured at fasted state (time = -60 min) during screening and both test visits (time = -60 min)
  C-Reactive Protein (CRP), assessed from blood samples at all visits
Markers of liver function | Measured at fasted state (time = -60 min) during screening and both test visits (time = -60 min)
  Concentrations of enzymes including but not limited to: Alanine Aminotransferase (ALAT), Aspartate Transaminase (ASAT).
Difference in self-reported energy intake | Measured 24-hours after test visits
  Difference in 24-h self-reported energy intake (E%) from carbohydrate, protein, and fat and total energy intake in response to the high carbohydrate vs. high protein isocaloric liquid meals.
Difference in energy intake from fat | Measured after meal consumption at t=150 min
  Difference in energy intake (E%) from protein during the ad libitum buffet in response to the high carbohydrate vs. high protein isocaloric liquid meals.
Difference in energy intake from protein | Measured after meal consumption at t=150 min
  Difference in energy intake (E%) from protein during the ad libitum buffet in response to the high carbohydrate vs. high protein isocaloric liquid meals.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas S Salling Quist, MSc, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No